CLINICAL TRIAL: NCT03651323
Title: Left Atrial Appendage Closure for Stroke Prevention in Atrial Fibrillation: Latin America Registry on WatchmanTM Outcomes in Real Life
Brief Title: Latin America Registry on WatchmanTM Outcomes in Real Life
Acronym: LATINAWERICA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Centro Medico Docente la Trinidad (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Luis Cressa, Interventional Cardiologist, Centro Medico Docente la Trinidad
Other Study IDs: ISRCAR00144
Record Dates: First submitted 2018-08-24; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Left atrial appendage; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Left atrial appendage closure with Watchman device — Percutaneous left atrial appendage closure using Watchman device

SUMMARY:
Left atrial appendage (LAA) occlusion with WatchmanTM has emerged as viable alternative to anticoagulation therapy in randomized controlled trials. The device has FDA approved since 2015 and the firsts Latin American cases were performed in 2012. However, there is no real world data from Latin American experience in terms of success and outcomes.

DETAILED DESCRIPTION:
Approximately 450 subjects will be enrolled in the study. Up to 50 sites in Latin America will participate in the study.

Primary analyses may include, but will not be limited to, the following: procedural complications, incidence of stroke and death. Descriptive statistics will be used for baseline, procedure and follow-up data collected through the registry.

Clinical history of each patient will be analyzed for a period of 6 months after the procedure according the standard practice at the enrolling centers. There will be no additional visits, nor procedures, for subjects in the registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were eligible for a WatchmanTM device implantation according to current international and local guidelines and per physician and institution discretion.

Exclusion Criteria:

* Patient who were currently enrolled in another investigational study or registry that would directly interfere with the current study aims.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation and indication for left atrial appendage closure
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Periprocedural complications | At implant
  Pericardial effusion, stroke, device embolization and bleeding
Incidence of Stroke | 6 months follow up
  Stroke
Incidence of Death | 6 months follow up
  Cardiovascular and no cardiovascular death

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Medico Docente la Trinidad, Caracas, Miranda, Venezuela

IPD SHARING:
Plan to Share IPD: No